CLINICAL TRIAL: NCT05224349
Title: Effectiveness and Safety of SMART BoNT-A Therapy With Dysport® in Patients With Post-stroke Chronic Upper Limb Spasticity in Real-life Setting.
Brief Title: Effectiveness and Safety of SMART [Spastic Muscle Palpation by Anatomic Landscape for BoNT-A (Botulinumtoxin-A) Injection to Reduce Muscle Tone] BoNT-A Therapy With Dysport® in Patients With Post-stroke Chronic Upper Limb Spasticity (ULS) in Real-life Setting.
Acronym: SMART-NIS
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-52120-456; EUPAS107722 (Other: EMA RWC)
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Post-Stroke Chronic Upper Limb Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Participants with stable oral anti-spasticity treatment for at least 4 weeks prior to study entry
- Group B: Participants with no anti-spasticity therapy for at least 4 weeks prior to study entry

SUMMARY:
The purpose of this study is to collect data for Dysport® SMART BoNT-A therapy usage in an office-based setting in post-stroke participants with chronic (> 6 months) focal Upper Limb Spasticity who have been under stable oral antispastics treatment or patients with no current anti-spasticity treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years with the capacity to consent.
* Subjects with a post-stroke medium to severe focal upper limb spasticity for at least 6 months. Medium to severe focal upper limb spasticity is defined as MAS ≥2 in the PTMG and DAS ≥2 in the PTT.
* Cohort according to SMART guidelines. The SMART injection concept is designed to be used only in patients suffering from simple patterns ("easy to diagnose spasticity pattern") of adult ULS, where Abobotulinumtoxin-A (AboBoNT-A) (Dysport®) injection can be simplified, by recognizing common spasticity patterns and key muscles for injection, identifying those muscles by palpation, and appropriate injection points of the suggested muscles using anatomic landmarks.
* Subjects with treatment goals as reduction of pain, reduction of muscle tone, improvement of care (hygiene/dressing) and/or improvement of passive motion.
* Subjects with the intention to be treated with Dysport® according to the current local Summary of Product Characteristics (SmPC) (Germany) and injection according to SMART must be taken prior to the entry in the study.
* Physiotherapy should remain unchanged within 4 weeks before study start.

Exclusion Criteria:

* Patients treated with intrathecal Baclofen or BoNT-A within the last 6 months
* If treated with oral spasticity medication, change of oral spasticity medication within the last 4 weeks
* Patients with active hand functions or patients with treatment goals of active functions.
* Patients with any contraindication for Dysport® according to SmPC.
* Patients in whom SMART therapy is not appropriate (e.g. spasticity pattern other than specified in SMART guidelines).
* Participation in an interventional trial at the same time and/or within 3 months before baseline.
* Diagnosed contracture/contracted muscle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with post-stroke chronic upper limb spasticity treated with Dysport® according to SMART guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Disability Assessment Scale (DAS) score in Principle Target of Treatment (PTT) for the upper limb. | At 12 weeks to 16 weeks after injection at Visit 1
  The PTT will be pre-selected from the 4 DAS domains: hygiene, dressing, limb position and pain of the upper limb at Visit 1. The extent of functional impairment in the PTT will be assessed on a four-point scale (range 0 to 3, where 0=no disability, and 3=severe disability) at each visit.

SECONDARY OUTCOMES:
Change from baseline of Modified Ashworth Scale (MAS) Primary Target Muscle Group (PTMG) | At 12 weeks to 16 weeks
  Muscle tone will be evaluated using the MAS. The PTMG (shoulder adductors, elbow flexors, wrist flexors or finger flexors) will be pre-selected at Visit 1. The muscle tone in the PTMG will be assessed from 0 (no increase in tone) to 4 (affected part(s) rigid in flexion or extension) at each visit.
Change from baseline of pain assessed with Visual Analogue Scale (VAS) | At 12 weeks to 16 weeks
  Pain (from 0 (no pain) to 10 (maximum pain) in upper limb extremity will be assessed at each visit.
Change from baseline of Spasticity Related Quality of Life Tool (SQoL-6D) | At 12 weeks to 16 weeks
  The questionnaire covers six dimensions: Pain/ discomfort, involuntary movement or spasms, restricted range of movement, caring for the affected limb, using the affected limb, mobility/balance. Each dimension is assessed using a five-point scale ranging from 0 to 4, with higher scores meaning worse outcome.
Incidence of Adverse Events (AEs) | Up to 32 weeks
Incidence of Special Situations (SS) | Up to 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (31):
- Germany (31):
  - Nervenarztpraxis, Altdorf
  - Neurologisches Zentrum, Berlin
  - Neurozentrum Erding, Erding
  - Praxis für Neurochirurgie und Schmerztherapie, Essen
  - Fürth; Medzentrum Fürth (MVZ), Fürth
  - Neuropraxis Fuerth, Fürth
  - Neuropraxis Fürth, Fürth
  - Evangelisches Klinikum Gelsenkirchen GmbH, Gelsenkirchen
  - Universitätsmedizin Greifswald, Greifswald
  - Herford; Klinikum Herford, Herford
  - Praxis Sojka-Raytscheff, Kiel
  - Neurologie am Funkerberg, Königs Wusterhausen
  - MVZ Lakumed gGMBH, Landshut
  - Praxis, Leipzig
  - Fuerth; Medzentrum Fuerth, Ludwigsburg
  - UK Schleswig-Holstein Campus Lübeck, Lübeck
  - Neuropraxis Mannheim, Mannheim
  - Neurozentrum Arabellapark, München
  - ABC Ambulantes BehandlungsCentrum GmbH, Nuremberg
  - ABC Moegeldorf, Nuremberg
  - Nürnberg; Praxis, Nuremberg
  - Gesundheitszentrum Quickborn, Quickborn
  - Medicum. Tegernsee, Rottach
  - Medicum. tegernsee - Rottach-Weissach, Rottach-Egern
  - ZNS Südpfalz, Rülzheim
  - St. Lukas Klinik GmbH, Solingen
  - Praxis, Sonneberg
  - Stadtroda; Asklepios Fachklinikum Stadtroda, Stadtroda
  - Gemeinschaftspraxis, Straubing
  - MVZ Neurologie am St. Johannes Sieglar, Troisdorf
  - Neurologie im Denkmal, Wuelfrath

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/